CLINICAL TRIAL: NCT06754202
Title: Silver Agri Age: Longevity, Intrinsic Capacity and Cognitive Impairment Into Farmlands and Natural Environments: Updating Contexts Following the "Montessori" Action
Acronym: Silver Agri Ag
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Collaborators: Regione Marche (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INRCA_005_2024
Record Dates: First submitted 2024-12-23; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: older people; mild cognitive impairment; social farming; montessori approach
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: pre-post study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects with mild cognitive impairment (MCI) (Experimental): Subjects with mild cognitive oimpairment (MCI) and self-sufficient in mobility that agreed to partecipate in various activities in rural enviroment.
  Interventions: Other: Social activities with cognitive stimulation

INTERVENTIONS:
Other: Social activities with cognitive stimulation — The nine-month program will include social activities following the "Montessori" action in the context of the agricultural multifunctionality such as horticulture, pet therapy, occupational therapy, sensory labs, physical activity held three days a week for five hours each day.

SUMMARY:
This project aims to enhance the intrinsic capacities of elderly individuals with mild cognitive impairment by promoting innovative activities based on the Montessori approach within the context of agricultural multifunctionality.

By selecting a rural environment with educational characteristics, we aim to involve individuals with mild cognitive deficits and their families in a personalized therapeutic journey. Through various activities, including horticulture, pet therapy, occupational therapies, sensory and food laboratories, we stimulate cognitive and motor skills, promoting a healthy and balanced lifestyle

DETAILED DESCRIPTION:
Promoting innovative activities following the "Montessori" action in the context of the agricultural multifunctionality, in order to leverage the intrinsic capacity in older people with cognitive impairment.

* Identifying a rural environment with educational features.
* Identifying individuals with mild cognitive impairments and relations with their families.
* Outlining individual therapeutic goals for each participant through different activities:

horticulture, pet therapy, occupational therapies, sensory laboratories, functional food laboratories for a healthy and balanced diet suitable for the first symptoms of dementia, physical activity and continuous social activity between different generations.

* Horticulture, pet therapy, occupational therapy, sensory labs, physical activity, and social activities IN CONTINUITY between different generations.
* Spreading the results to a wide National and International audience.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild cognitive impairment (MCI);
* Mini Mental State Examination ≥ 24;
* ability and willingness to sign informed consent

Exclusion Criteria:

* Mini Mental State Examination < 24;
* severe visual impairment;
* inability to walk without help or assistance, Tinetti's scale <20

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-03 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in the positive and negative affects | At baseline and after 9 months
  The PANAS (Positive and Negative Affect Schedule) produces two distinct dimensions of affect: Positive Affect (PA): Measures emotions like joy, interest, excitement, and enthusiasm and Negative Affect (NA): Measures emotions like fear, anger, sadness, and guilt. Participants rate each of the 20 items (10 for PA, 10 for NA) on a 5-point scale (from 1 = "Very slightly or not at all" to 5 = "Extremely"). The possible score range for both PA and NA is 10 to 50.
  Higher scores indicate higher levels of that particular affect Scores for each subscale are calculated by summing the ratings for the corresponding items.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gagliardi, MsC, Study Chair — IRCCS INRCA
Locations (2):
- Italy (2):
  - INRCA Hospital, Ancona
  - INRCA Hospital, Fermo

REFERENCES:
- [Derived] Gambella E, Lombardi L, Cicconi D, Raccichini A, Paciaroni L, Giuli C, Bonfigli AR, Fabbietti P, Pelliccioni G, Gagliardi C. The Silver Agri Age project in Italy: a Montessori-inspired social intervention with older adults with mild cognitive impairment. Single-group pre-post pilot study protocol. Front Public Health. 2025 May 16;13:1561263. doi: 10.3389/fpubh.2025.1561263. eCollection 2025. PMID 40453497